CLINICAL TRIAL: NCT02776241
Title: Effect of Water Intake and Water Restriction on Total Kidney Volume in Autosomal Dominant Polycystic Kidney: The HYDRA Study
Brief Title: Effect of Water Intake and Water Restriction on Total Kidney Volume in Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Signe Vinsand Naver, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HYDRA
Record Dates: First submitted 2016-05-04; First posted 2016-05-18 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: ADPKD
Keywords: ADPKD; total kidney volume; kidney disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- water restriction (No Intervention): 20 patients will be subjected to 3 hours of water restriction following MR scan of the kidneys.
- high water intake (Active Comparator): 20 patients will be subjected to 1 hour of high water intake (20 ml/kg) following MR scan of the kidneys.
  Interventions: Other: water

INTERVENTIONS:
Other: water
  Arms: high water intake

SUMMARY:
The objective of this study is to measure the influence of both short term water restriction and high water intake on total kidney volume, measured by Magnetic Resonance Imaging (MRI) scan in Autosomal Dominant Polycystic Kidney Disease (ADPKD) patients.

DETAILED DESCRIPTION:
Patients will be randomized to either water restriction for 3 hours or high water intake (20 ml/kg) for 1 hour. Before intervention and after intervention patients will have an MRI scan of the kidneys to measure the total kidney volume (TKV) (differentiated in cortex, medulla and cyst volume). The objective is to identify whether water restriction or high water load will change the TKV. Secondly investigators will analyze different biomarkers (aldosterone, renin, vasopressin/copeptin, urine- and blood-osmolarity) before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD
* CKD stage 1-3

Exclusion Criteria:

* Patients treated with diuretics
* Pregnancy
* Change in antihypertensive treatment < 1 month
* Any condition contraindicating MR scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in total kidney volume | Baseline and 3 hours

SECONDARY OUTCOMES:
Change in total cyst volume | Baseline and 3 hours
Change in plasma renin | Baseline and 3 hours
Change in plasma aldosterone | Baseline and 3 hours
Change in plasma copeptin | Baseline and 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Signe V Naver, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes